CLINICAL TRIAL: NCT01606449
Title: Thirty-year Follow-up of a Case Series of Patients Operated Upon for Type II-IV Hiatal Hernia
Brief Title: Follow-up of Patients Operated Upon for Type II-IV Hiatal Hernia
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Sandro Mattioli, Associate Professor M.D., University of Bologna
Other Study IDs: UniBoDipTrap2; II-IV HH (Registry Identifier: Type II-IV Hiatal Hernia)
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-01

CONDITIONS: Gastroesophageal Reflux Disease With Hiatal Hernia; Paraesophageal Hernia
Keywords: Gastroesophageal reflux diseases; Hiatal Hernia; Paraesophageal Hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Group 1 = Patients with type II Hiatal Hernia submitted to surgical therapy
  Interventions: Procedure: Surgical Therapy
- Group 2: Group 2 = Patients with type III Hiatal Hernia submitted to surgical therapy
  Interventions: Procedure: Surgical Therapy
- Group 3: Group 3 = Patients with type IV Hiatal Hernia submitted to surgical therapy
  Interventions: Procedure: Surgical Therapy

INTERVENTIONS:
Procedure: Surgical Therapy — Open Anti-reflux fundoplication according to Nissen-Rossetti, floppy Nissen, Belsey MK IV,Collis Nissen, Collis-Belsey.
  Minimally-Invasive fundoplication according to floppy Nissen, left thoracoscopic Collis-laparoscopic Nissen.

SUMMARY:
Surgical therapy for gastroesophageal reflux disease (GERD) and hiatal hernia (HH) can achieve outcomes that afford the patient lifelong satisfaction. The published results obtained with this surgery may not be considered to be definitive in relation to the length of follow-up or patients' life expectancy. The real recurrence rates and the results of surgery for GERD are difficult to assess due to the lack of serial time points during the follow-up. Further bias may have been introduced into the analysis by a lack of appropriate controls. The results of surgical therapy for type II-IV HH are even more controversial because of the high rate of anatomical relapse and the different methods of follow-up adopted in reported case series.

Aim of this study is to clarify the value of surgical therapy for type II-IV HH. The investigators report on patients who were followed up after surgery at various time points over the course of 30 years.

DETAILED DESCRIPTION:
We reviewed the charts of patients who underwent primary surgery for type II-IV Hiatal Hernia during the period from January 1980 - December 2010.

Pre-operatively, the patients routinely underwent symptom assessment, a barium swallow, upper GI endoscopy and esophageal manometry.

The principles of surgery for GERD and hiatal hernias involve full isolation of the diaphragmatic pillars and E-G junction, full isolation and resection of the sac and fat pad into the mediastinum (except for the fat close to the lesser curvature, to preserve the integrity of the vagus nerves), evaluation of the degree of esophageal shortening, and a Collis gastroplasty in cases of short esophagi.

Post-operatively, the patients participated in a free-of-charge outpatient follow-up program at 6 months, 12 months and every year for 5 years.

The length of the follow-up was calculated from the day of the surgery to the day that the patient underwent the last complete follow-up. The type and severity of symptoms and the grade of reflux esophagitis were scored using a questionnaire with semi-quantitative scales (from 0 = absence of symptoms and esophagitis to 3 = severe symptoms and esophagitis). An evaluation scale for the surgical results, with scores ranging from "excellent" to "poor", was also used.

ELIGIBILITY:
Inclusion Criteria:

* patients aged > 18 years, undergoing surgery for the treatment of type II-IV hiatal hernia ± GERD.

Exclusion Criteria:

* association of GERD with epiphrenic esophageal diverticulum
* collagen diseases
* undetermined esophageal motility disorders, redo antireflux surgery
* previous surgery on the thoracic and abdominal esophagus and stomach, on the diaphragm.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consecutively operated upon for type II-IV hiatal hernia in the period January 1980-December 2010.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 1980-01; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Mattioli, MD, Principal Investigator — Department of General Surgery and Organ Transplantations
Locations (1):
- Department of General Surgery and Organ Transplantation, Bologna, Italy

REFERENCES:
- [Derived] Lugaresi M, Mattioli B, Daddi N, Di Simone MP, Perrone O, Mattioli S. Surgery for Type III-IV hiatal hernia: anatomical recurrence and global results after elective treatment of short oesophagus with open and minimally invasive surgery. Eur J Cardiothorac Surg. 2016 Apr;49(4):1137-43. doi: 10.1093/ejcts/ezv280. Epub 2015 Sep 16. PMID 26377635